CLINICAL TRIAL: NCT02817646
Title: A Retrospective Investigator Initiated Trial Evaluating Protein Intake and CT Assessments of Muscle Mass of Critically Ill Patients in Relation to Outcome Parameters: the PROMUS-study
Brief Title: Study in ICU Patients Regarding Protein Intake and CT-derived Body Composition
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Wilhelmus G.P.M. Looijaard, MD, PhD Candidate, Amsterdam UMC, location VUmc
Other Study IDs: ICUPROMUS
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Muscular Atrophy
Keywords: Intensive Care Unit; Critical Illness; Body composition; Protein nutrition
MeSH Terms: conditions — Muscular Atrophy; Critical Illness | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intensive care patients: Patients admitted to the intensive care unit for 4 days or more with a computed tomography scan made for clinical reasons early during intensive care stay and who receive enteral and/or parenteral nutrition as per hospital protocol
  Interventions: Other: Computed tomography scan made for clinical reasons; Dietary Supplement: Nutrition as per hospital protocol

INTERVENTIONS:
Other: Computed tomography scan made for clinical reasons — Patients were included if a computed tomography scan of the abdomen or thorax was made early during intensive care admission (1 day before up to 4 days after admission)
Dietary Supplement: Nutrition as per hospital protocol — Patients received enteral and/or parenteral nutrition as per usual hospital protocol

SUMMARY:
The purpose of this study is to determine whether protein intake during the first days of intensive care admission, in relation to body composition at intensive care admission as assessed on computed tomography scans made during routine care, is are related to clinical outcome in critically ill patients.

DETAILED DESCRIPTION:
Optimal protein and energy intake have been shown to be relevant for reducing mortality in prospective observational studies in mechanically ventilated patients admitted to the intensive care unit. However, nutritional status (protein mass, muscle mass) of patients at admission and possible consequences for clinical outcome are largely unknown. Computerized tomography scans can be used to assess muscle mass as a proxy for body protein mass.

The investigators are especially interested in the effect of protein intake on clinical outcome in intensive care patients with different body protein mass at admission. This is relevant for appropriate formulation of clinical (protein) nutrition in this patient group. Therefore, the relationship between protein intake and patient outcome is evaluated in intensive care patients with low muscle and normal muscle area, using muscle area from computed tomography scans as a proxy of body protein mass.

Additionally, data from computed tomography scans regarding muscle quality and muscle- and fat quantity are used to evaluate the prognostic value of body composition at intensive care admission. Finally, abdominal computed tomography scans are compared with thoracic computed tomography scans.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal computed tomography scan made 1 day before up to 4 days after admission to the intensive care unit
* Length of intensive care stay of at least 4 days
* Mechanical ventilation during intensive care stay

Exclusion Criteria:

* Computed tomography scan not eligible for analysis
* Missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-02; Primary Completion 2016-10 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 6-months after intensive care admission
All-cause mortality | 28-days after intensive care admission
All-cause mortality | 60-days after intensive care admission
All-cause mortality | 90-days after intensive care admission
All-cause mortality | From admission to the intensive care unit untill discharge from the intensive care unit, an average of two weeks
All-cause mortality | From admission to the intensive care unit untill discharge from the hospital, an average of one month

SECONDARY OUTCOMES:
Percentage of patients discharged to home | After discharge from the hospital, on average after one month
Length of hospital stay (days) | The total duration of admission to the hospital, an average of one month
Length of intensive care unit stay | The total duration of admission to the intensive care unit, an average of two weeks
Length of ventilation | The total duration of mechanical ventilation during intensive care unit stay, an average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Weijs, PhD, Study Director — Amsterdam UMC, location VUmc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weijs PJ, Looijaard WG, Beishuizen A, Girbes AR, Oudemans-van Straaten HM. Early high protein intake is associated with low mortality and energy overfeeding with high mortality in non-septic mechanically ventilated critically ill patients. Crit Care. 2014 Dec 14;18(6):701. doi: 10.1186/s13054-014-0701-z. PMID 25499096
- [Result] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Result] Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Twisk JW, Oudemans-van Straaten HM, Weijs PJ. Skeletal muscle quality as assessed by CT-derived skeletal muscle density is associated with 6-month mortality in mechanically ventilated critically ill patients. Crit Care. 2016 Dec 1;20(1):386. doi: 10.1186/s13054-016-1563-3. PMID 27903267